CLINICAL TRIAL: NCT00351572
Title: Frequency of Circulating Tumour Cells in Stage II and Stage III Colon Cancer Patients
Status: Completed | Type: Observational
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: GI-5-0055
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Colon Cancer
Keywords: colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Cell Search Assay

SUMMARY:
This study will determine whether a new diagnostic test called the Cell Search Assay can detect circulating colon cancer cells in patients who have had surgery for colon cancer and had visible cancer removed. Other parts of the study will look at whether the presence of the circulating tumor cells in blood predicts whether a patient will have their colon cancer return.

ELIGIBILITY:
Inclusion Criteria:

* stage II or III colon cancer

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic and any other interested parties
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada